CLINICAL TRIAL: NCT04828512
Title: Subclinical Diabetes Confirmed by 75gm-OGTT Influence on the Prognosis of Decompensated Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: CR 313032
Record Dates: First submitted 2021-03-22; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 42 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal glucose tolerance (NGT): In the 75-g OGTT, an FPG level of < 100 mg/dL or a 120-min PG level of < 140 was diagnosed as NGT.
- impaired glucose intolerance (IGT): In the 75-g OGTT, an FPG level of 100-125 mg/dL (5.6-6.9 mmol/L) or a 120-min PG level of 140-200 mg/dL (7.8-11.1 mmol/L) was diagnosed as IGT.
- newly diagnosed DM (subclinical DM): In the 75-g OGTT, a basal FPG level ˃126 mg/dL (7.0 mmol/L) or a 120-min PG level ˃200 mg/dL (11.1 mmol/L) was considered as newly diagnosed DM (hereafter referred to as subclinical DM).

SUMMARY:
Disorders of glucose metabolism, such as impaired glucose intolerance (IGT) and diabetes mellitus (DM), frequently occur in cirrhosis. However, it has been underestimated when fasting plasma glucose (FPG) levels are considered. We aimed to evaluate who needs to be undertaken a 75-g oral glucose tolerance test (OGTT) to find underlying subclinical diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Admitted to a hospital

Exclusion Criteria:

* Previously confirmed DM
* Being treated for DM
* Standard risk factors of T2DM, such as high body mass index and family history of diabetes
* Symptoms of DM, such as increased thirst and the need to urinate
* Either hepatocellular carcinoma or other malignancy
* Hepatic failure or uncontrolled decompensation [that is, refractory ascites or active variceal hemorrhage]
* Significant illnesses such as sepsis that may have interfered with glucose metabolism
* Pancreatic dysfunction such as acute/chronic pancreatitis that may have affected glucose metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cirrhosis without previous diabetes history
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2007-01-02 (Actual); Primary Completion 2014-01-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival | through study completion, an average of 3 year
  Overall survival

SECONDARY OUTCOMES:
major complications of cirrhosis | through study completion, an average of 3 year
  hepatic encephalopathy (HE), the development of spontaneous bacterial peritonitis (SBP), acute kidney injury (AKI), variceal bleeding, and infection

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang SH, Kim MY, Han SK, Baik SK. Subclinical diabetes confirmed by 75-g OGTT influence on the prognosis of decompensated cirrhosis. J Gastroenterol Hepatol. 2024 Jan;39(1):172-179. doi: 10.1111/jgh.16327. Epub 2023 Sep 11. PMID 37697655